CLINICAL TRIAL: NCT04368520
Title: Clinical Trial to Optimise Levels of Vitamin D for Rhinovirus Protection (COLD)
Brief Title: Clinical Trial to Optimise Levels of Vitamin D for Rhinovirus Protection
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID-19 pandemic prevented start-up
Sponsor: Queen Mary University of London (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: COLDstudy
Record Dates: First submitted 2020-03-26; First posted 2020-04-29 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Common Cold
Keywords: Rhinovirus
MeSH Terms: conditions — Common Cold | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Two treatment arms of vitamin D3: low dose (800IU) vs. high dose (3,200IU) given daily, for 3 months
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Low dose vitamin D3 (Experimental)
  Interventions: Dietary Supplement: Vitamin D3
- High dose vitamin D3 (Experimental)
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 800 IU Fultium-D3, cholecalciferol (Internis), given daily for 3 months
  Arms: Low dose vitamin D3
Dietary Supplement: Vitamin D3 — 3,200 IU Fultium-D3, cholecalciferol (Internis), given daily for 3 months
  Arms: High dose vitamin D3
Other: Placebo — Hypromellose capsules, given daily for 3 months
  Arms: Placebo

SUMMARY:
A phase II randomised, placebo-controlled trial to identify the optimal regimen of vitamin D supplementation for rhinovirus protection, determined by host responses to a clinically induced rhinovirus challenge. The primary outcome is rhinovirus titre after inoculation with rhinovirus; secondary outcomes are self-reported respiratory symptom scores, concentrations of cytokines and chemokines sampled from the nasal mucosa, and the transcriptional responses of nasal epithelial cells.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years
2. Gives written informed consent
3. Serum 25-hydroxyvitamin D concentration <75 nmol/L
4. Agrees not to take supplement containing vitamin D during participation
5. Agrees not to commence smoking or vaping during participation

Exclusion criteria:

1. Current smoker or vaper
2. Taken vitamin D supplement or other supplement containing vitamin D, in previous 3 months
3. Sunny holiday abroadI, defined as any location 51 degrees North/South of the equator, for ≥1 week, in the previous 3 months
4. Dependent(s) <6 months old
5. Positive serology for anti-RV16 antibodies
6. Living with someone with severe airways disease
7. Any of the following medical conditions:

   1. Diabetes mellitus
   2. Asthma
   3. Chronic Obstructive Pulmonary Disease
   4. Respiratory allergies
   5. Sarcoidosis
   6. Hyperparathyroidism
   7. Nephrolithiasis
   8. Active tuberculosis
   9. Liver failure
   10. Renal failure
   11. Lymphoma or other malignancy not in remission for ≥ 3 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Rhinovirus titres | +3 to +5 days after inoculation
  PCR-detected rhinovirus-16 load sampled from the nasal mucosa

SECONDARY OUTCOMES:
Respiratory symptom score (Jackson Score) | +1 to +14 days after inoculation
  Total self-reported respiratory symptom score (scored 0-32; increasing score equals increasing symptom severity)
Cytokine and chemokine concentrations | Day 0 and +4 days after inoculation
  Change in concentrations of inflammatory mediators (Including, but not limited to IL-1β, IL-2, IL-4, IL-5, Il-6, IL- 7, IL-8 [CXCL8], IL-10, IL-12, IL-13, IL-15, IL-17, IL-1RA, IL-2R, IFN-α, IFN-γ, TNF-α, MCP-1 [CCL2], MIP- 1α [CCL3], MIP-1β [CCL4], RANTES [CCL5], eotaxin [CCL11], MIG [CXCL9], IP-10 [CXCL10], EGF, FGF-basic, HGF, VEGF, G-CSF, GM-CSF)
Change in level of vitamin D-regulated gene expression | Day 0 and +4 days after inoculation
  Change in expression of DHCR7, CYP2R1, CYP3A4, CYP27A1, CYP27B1, CYP24A1, VDR, DBP, RXRA

CONTACTS AND LOCATIONS:
Locations (1):
- St. Mary's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be shared with other researchers subject to terms of Data Transfer Agreement and IRB approval
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 2 years after completion of the trial